CLINICAL TRIAL: NCT02571712
Title: Evaluation of the Safety of GANFORT® (Bimatoprost 0.03% Plus Timolol 0.5%) Ophthalmic Solution in Chinese Patients With Open-angle Glaucoma or Ocular Hypertension
Brief Title: Safety of GANFORT® Ophthalmic Solution in Chinese Patients With Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 192024-094
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Ganfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GANFORT® (Other): One drop of GANFORT® (bimatoprost 0.03% plus timolol 0.5%) instilled in each affected eye once daily in the evening for 24 weeks.
  Interventions: Drug: bimatoprost 0.03% plus timolol 0.5%

INTERVENTIONS:
Drug: bimatoprost 0.03% plus timolol 0.5% — 1 drop of bimatoprost 0.03% plus timolol 0.5% (GANFORT®) instilled in the affected eye once daily.
  Other Names: GANFORT®

SUMMARY:
A study to evaluate the long-term safety of GANFORT® (bimatoprost 0.03% plus timolol 0.5%) in Chinese patients with open-angle glaucoma or ocular hypertension who are insufficiently responsive to topical beta-blocker or prostaglandin analogues.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension that is insufficiently responsive to topical beta-blockers or prostaglandin analogues in one or both eyes
* Is willing to stop other intraocular pressure (IOP)-lowering medications and switch to GANFORT® as a single agent in affected eye(s).

Exclusion Criteria:

* Reactive airway disease including bronchial asthma or a history of bronchial asthma or severe chronic obstructive pulmonary disease
* Sinus bradycardia, sick sinus syndrome, sino-atrial block, second or third degree atrioventricular block, not controlled with pacemaker. Overt cardiac failure, cardiogenic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne McLaughlin, Study Director — Allergan
Locations (15):
- China (15):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tongren hospital Capital Medical University, Beijing, Beijing Municipality
  - Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Eye Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Henan Provincial Eye Hospital, Henan, Zhengzhou

REFERENCES:
- [Derived] Sun X, Yao K, Liu Q, Zhang H, Xing X, Fang A, Duan X, Yu M, Chen MY, Yang J, Goodkin ML. Safety of Fixed-Combination Bimatoprost 0.03%/Timolol 0.5% Ophthalmic Solution at 6 Months in Chinese Patients with Open-Angle Glaucoma or Ocular Hypertension. Ophthalmol Ther. 2023 Feb;12(1):341-353. doi: 10.1007/s40123-022-00593-w. Epub 2022 Nov 12. PMID 36370233
- See also: More Information — http://www.allerganclinicaltrials.com